CLINICAL TRIAL: NCT04870229
Title: Carnosine for Peripheral Arterial Disease (Car-PAD)
Brief Title: Carnosine for Peripheral Arterial Disease
Acronym: (Car-PAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Shahid Baba, Assistant Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16.0047
Record Dates: First submitted 2019-07-17; First posted 2021-05-03 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Carnosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Carnosine (Active Comparator): Each participant will be given a daily oral dose 1g of methycellulose powder for 6 months
  Interventions: Drug: Carnosine
- Placebo (Placebo Comparator): Each participant will be given a daily oral dose 1g of placebo for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carnosine
  Arms: Carnosine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The hypothesis is that oral supplementation of L-carnosine will inhibit PHDs, increase HIF1-translocation and angiogenesis and thus improve the functioning of lower extremities in PAD patients.

Primary Aim:

1. Compare the effect of carnosine and placebo supplementation on the 6MWT in PAD patients with and without claudication.

Secondary Aim:

1. Determine whether carnosine supplementation improves the pain-free treadmill walking ability of the subjects supplemented with carnosine compared to placebo.
2. Compare the levels of carnosine, VEGF, HIF-1α, and PHDs activity in the skeletal muscle before and after placebo and carnosine supplementation.
3. Compare the levels of EPCs (CD34+/CD133+), inflammatory markers (serum amyloid A, hsCRP) and thrombotic markers (fibrinogen, homocysteine) as cardiovascular risk markers in these subjects.
4. Explore the effects of race and gender on VEG, carnosine, and HIF-1α levels in both groups.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is caused by atherosclerotic occlusion of the lower extremities that reduces blood flow and leads to intermittent claudication and critical limb ischemia. PAD is diagnosed by calculating the ratio of blood pressure at the ankle to that of the arm (the ankle-brachial index [ABI]). An ABI of <0.90 is indicative of atherosclerosis in the leg. Recent data from developed and developing countries have estimated that >200 million people worldwide and approximately 12 million people in United States have PAD. Both symptomatic and asymptomatic PAD patients have an increased risk of mortality, morbidity, and a lower quality of life. With the increasing incidence of type 2 diabetes (T2D) and a rising aging population, the number of PAD patients is likely to increase. Because PAD is an under-recognized disease, currently few medications are available to improve the functional performance of these patients. Although surgical revascularization is an available treatment, grafts can fail and the stenosis can reoccur in these patients.

To adequately compensate the loss of tissue due to occlusion, the current emphasis is to increase the therapeutic angiogenesis and arteriogenesis in the ischemic limb that could improve the walking ability and the quality of life in PAD patients. Pre-clinical studies have shown that supplementation of carnosine (500 mg/day) in heart failure patients for 6 months improves their performance on the 6-minute walking test (6MWT) compared with placebo-treated patients. Similarly supplementation of carnosine (2g/day) for 12 weeks has been shown to normalize glucose intolerance and reduce insulin levels in obese individuals. No side effects were reported at these doses. Carnosine (β-alanine-histidine) is a histidyl dipeptide present in high concentration in the skeletal muscle, brain, and heart. It is a food constituent that is present in red meat, chicken, and turkey. This dipeptide is synthesized by the ATP grasp enzyme carnosine synthetase6 and hydrolyzed to β-alanine and histidine by the serum and kidney carnosinase. Carnosine has the abilities to quench reactive aldehydes, bind metals, and buffer intracellular pH. Numerous studies have shown that the supplementation of -alanine increases the levels of carnosine in the skeletal muscle and improves the exercise performance in humans. Our preliminary studies with the mice model of hind limb ischemia (HLI) shows that both the pretreatment and the supplementation of carnosine after femoral artery ligation increases blood flow in the ischemic limb compared with the non-treated mice. Mechanistic studies show that the supplementation of carnosine increases angiogenic factor VEGF and endothelial progenitor cells mobilization in the carnosine treated HLI mice. Similarly the stabilization of HIF-1α, the master regulator of angiogenesis and angiogenic factor VEGF, is increased in the hypoxic C2C12 cells (murine myoblasts).

Based on these pre-clinical studies and our initial observations the Investigator will examine whether supplementation of carnosine (1 g/day) to PAD patients for 6 months will improve walking performance compared with the placebo-treated patients. Further, the Investigator will examine whether the supplementation of carnosine increases the capacity of pain-free treadmill walking time and levels of VEGF, HIF-1α, and carnosine in the skeletal muscle of PAD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 50 and 80 years of age.
2. English Speaking.
3. ABI 0.3 -<0.90 (in at least one leg).
4. Willing to comply with protocol requirements.
5. Able to provide informed consent.
6. Able to walk on a treadmill for more than 2 minutes -

Exclusion Criteria:

1. Subjects with HIV, hepatitis, significant liver disease, active infection, anemia, organ transplant, renal disease requiring dialysis, lung disease requiring oxygen, significant congenital heart disease, cancer of any type, and untreated thyroid disease.
2. Diagnosis of carnosinemia.
3. Known allergy to L-carnosine or meat.
4. Obesity from a known genetic defect.
5. Dementia.
6. Critical limb ischemia with below or above knee amputations.
7. Foot ulcers.
8. Major amputations.
9. Participating in other clinical trials.
10. End stage renal disease.
11. Presence of significant injury within 30 days before enrollment.
12. Prisoners
13. Poorly controlled diabetes (HbA1C >9%).
14. Able to walk for more than 12 minutes.
15. Currently taking Pletal (cilostazol) or Trentol (pentoxifylline) -

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Walking Endurance | 6 months
  Compare effects of carnosine and placebo supplementation on the 6MWT in patient with and without claudication

SECONDARY OUTCOMES:
Graded treadmill test | 6 months
  We will measure the onset of claudication onset time and peak walk time

CONTACTS AND LOCATIONS:
Overall Officials: Shahid P Baba, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No